CLINICAL TRIAL: NCT02993809
Title: Autologous Transplantation of BM-ECs With Platelet-Rich Plasma Extract for the Treatment of Critical Limb Ischemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMEC-PRPE
Record Dates: First submitted 2016-11-23; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-09

CONDITIONS: Leg Ulcer; Diabetic Foot; Gangrene; Peripheral Vascular Disease; Ischemia
MeSH Terms: conditions — Leg Ulcer; Diabetic Foot; Gangrene; Peripheral Vascular Diseases; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BM-ECs and PRPE (Experimental): Multipoint of intramuscular injections into ischemic limbs.Injections composed of bone marrow derived endothelial cells (BM-ECs) and platelet-rich plasma extract (PRPE).
  Interventions: Biological: BM-ECs and PRPE
- BM-ECs (Active Comparator): Intramuscular injection of bone marrow derived endothelial cells only.
  Interventions: Biological: BM-ECs

INTERVENTIONS:
Biological: BM-ECs and PRPE
  Arms: BM-ECs and PRPE
Biological: BM-ECs
  Arms: BM-ECs

SUMMARY:
The intent of this clinical study is to evaluate the safety of the injection composed of autologous bone marrow derived endothelial cells (BM-ECs) and platelet-rich plasma extract (PRPE) for the treatment of critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

Limb ischemia patients(e.g. arteriosclerosis obliterans,diabetic critical limb ischemia, thromboangitis obliterans)

1. 18 Years to 80 Years (Adult, Senior);
2. Have ability to understand and comply with the study requirements, and provide the written informed consent prior to any procedures ;
3. Patient meets at least one of the following diagnostic criteria for the index limb:

   1. ABI<0.7mmHg
   2. TcpO2 <40 mm Hg
   3. Or, nonhealing ulcer due to local arterial compromise with no opportunity for revascularization;
4. Have no improvement after conservative treatment and are not suitable for surgical bypass surgery because no outflow tract of diseased vessel can be found by imaging;
5. Despite having good outflow artery, but the elderly and frail patients can also not tolerate revascularization or interventional surgery;
6. Unlikelihood of major amputation of the leg during the next 12 months;
7. Expected life span more than 2 years.

Exclusion Criteria:

1. Pregnant or lactating;
2. Diabetics with poorly controlled blood glucose levels (defined as HbA1c>7% and/or proliferative retinopathy);
3. Patients with decompensated cardiac, renal or liver disease;
4. Patients with confirmed malignant tumor;
5. Subjects are with serious heart, liver, kidney and lung failure or under poor general condition that are inability to undergo bone marrow harvesting and transplantation;
6. Known or suspected disease of the immune system or osteomyelitis;
7. Inability to sign informed consent form and to comply with the schedule of the study;
8. There has reason to suspect that the patient is forced to join the study;
9. Any other condition, in the opinion of the investigator, would render the patient unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Survival without major amputation | 6 months after implantation

SECONDARY OUTCOMES:
Perfusion rate in treated tissue by measure of ankle-brachial index (ABI) | Within 6 months after implantation
Perfusion rate in treated tissue by transcutaneous PO2 (TcPO2) | Within 6 months after implantation
Perfusion rate in treated tissue by digital subtraction angiography (DSA) | Within 6 months after implantation
wound size | Within 6 months after implantation
wound stage | Within 6 months after implantation
Pain intensity | Within 6 months after implantation
  Pain intensity using Visual Analogue Scale
Thermography | Within 6 months after implantation

IPD SHARING:
Plan to Share IPD: Yes